CLINICAL TRIAL: NCT07237464
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of GB18 Following Single Subcutaneous Injection in Healthy Adult Participants
Brief Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of GB18 Injection in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KXZY-GB18-101
Record Dates: First submitted 2025-09-26; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Cancer Cachexia (CC); Cancer Cachexia; Cancer Cachexia Syndrome
Keywords: Cancer cachexia; GB18; healthy adult; Phase I; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — alkaloid GB18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study and thus the Investigator, Sponsor, Sponsor's delegates (if applicable), and participants are all blinded to treatments. No individual participant information that can be potentially unblinded for the Investigator or participant will be reported until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- A1-50mg-GB18 (Experimental)
  Interventions: Drug: GB18 injection
- A1-50mg-placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- A2-100mg-GB18 (Experimental)
  Interventions: Drug: GB18 injection
- A2-100mg-placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- A3-200mg-GB18 (Experimental)
  Interventions: Drug: GB18 injection
- A3-200mg-placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- A4-400mg-GB18 (Experimental)
  Interventions: Drug: GB18 injection
- A4-400mg-placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- A5-600mg-GB18 (Experimental)
  Interventions: Drug: GB18 injection
- A5-600mg-placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB18 injection — GB18 will be administered to participants at a starting dose of 50 mg and increasing to 100, 200, 400 and 600 mg in sequential dosing cohorts.
  Arms: A1-50mg-GB18; A2-100mg-GB18; A3-200mg-GB18; A4-400mg-GB18; A5-600mg-GB18
Drug: Placebo — Placebo will be administered to participants at doses matching GB18.
  Arms: A1-50mg-placebo; A2-100mg-placebo; A3-200mg-placebo; A4-400mg-placebo; A5-600mg-placebo

SUMMARY:
This study is a first-in-human, randomized, double-blind, placebo-controlled, dose-escalation trial in healthy adult participants to evaluate the safety, tolerability, PK, PD, and immunogenicity of GB18.

A total of 36 healthy participants will be enrolled, including 5 dose cohorts (A1-A5) of 50 mg, 100 mg, 200 mg, 400 mg and 600 mg, with 4 participants in Cohort A1, and 8 participants per following cohorts (A2-A5). Participants in each cohort will be randomized to receive GB18 or placebo.

The arms of this study include:

To evaluate the safety and tolerability of GB18 following a single subcutaneous (SC) administered dose in healthy adult participants.

To characterize the serum pharmacokinetics (PK) of GB18 following a single SC administered dose in healthy adult participants.

To characterize the pharmacodynamics (PD) of a single SC administration of GB18 on circulating GDF15 concentrations in healthy adult participants.

To evaluate the immunogenicity profile of GB18 in healthy adult participants. To evaluate the effect of GB18 on body weight in healthy adult participants. To preliminary evaluation of the relationship between GB18 serum concentration and QTc interval after a single SC administration in healthy adult participants.

DETAILED DESCRIPTION:
This study is a first-in-human, randomized, double-blind, placebo-controlled, dose-escalation trial in healthy adult participants to evaluate the safety, tolerability, PK, PD, and immunogenicity of GB18.

A total of 36 healthy participants will be enrolled, including 5 dose cohorts (A1-A5) of 50 mg, 100 mg, 200 mg, 400 mg and 600 mg, with 4 participants in Cohort A1, and 8 participants per following cohorts (A2-A5). Participants in each cohort will be randomized to receive GB18 or placebo at a ratio of 3:1, with 3 participants receiving GB18 and 1 participant receiving placebo in Cohort A1, and 6 participants receiving GB18 and 2 participants receiving placebo in the remaining cohorts (A2-A5).

Healthy participants will be screened within 28 days prior to dosing. Participants will be admitted to the Clinical Research Unit (CRU) on Day -1 and receive a single subcutaneous dose of GB18 or placebo on Day 1 at the abdomen. Participants will receive safety assessments on Day 8 and can be discharged with the permission of the investigator. Safety assessments and PK/PD/immunogenicity sampling will be carried out at scheduled timepoints.

The participants will return to the CRU on Day 10, 15, 29, 50, 71, 92, 106 and 127 for blood sampling, safety, and other assessments such as vital signs, ECG, and laboratory test etc.

GB18 will be administered to participants at a starting dose of 50 mg and increasing to 100, 200, 400 and 600 mg in sequential dosing cohorts. The Safety Review Committee (SRC) will assess the safety data, PK data and available PD data at least up to Day 15 (Cohort A1-2)/29 (Cohort A3-5) after the dose administration of each cohort, and a decision of whether to escalate to the next higher dose level or adjust the dose or discontinue dosing will be made by the SRC.

For the safety of participants, 2 sentinel participants will be randomly dosed (GB18: placebo=1:1) at least 24 hours before the remaining participants in the cohort receive dosing, except for Cohort A1. Once safety is confirmed, the remaining participants will be dosed.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have signed the informed consent form (ICF) prior to the study, fully understand the content, procedures, and possible adverse reactions of the study, and are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
2. Male and female participants aged 18-55 years (inclusive), at the time of signing the ICF.
3. Body weight ≥ 50 kg for males and ≥ 45 kg for females, with a body mass index (BMI = weight (kg)/height 2 (m) 2) of 18.5-26 kg/m2 (inclusive).
4. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, Vital signs, 12-lead ECG, and laboratory tests.
5. Participants (including their partners) who have no plan to become pregnant and voluntarily use effective contraception from screening to 6 months after the last dose.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of HIV infection, syphilis, hepatitis B, or hepatitis C; positive testing for HIV, syphilis, HBsAg, or HCVAb.
3. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody or molecules made of components of monoclonal antibodies.
4. History of recurrent infections or active infections.
5. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior, or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. Smoking more than five cigarettes per day on average, or habitually used nicotine containing products, or unable to refrain from smoking during the trial.
7. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
8. Exposure to live vaccines within 28 days of screening.
9. Previous administration with an investigational drug within 30 days or marketed or investigational monoclonal antibodies within 3 months or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
10. History of drug abuse within the past 5 years or use of drugs in the 3 months prior to screening, or a positive urine drug test at screening.
11. Screening BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
12. Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, or QRS interval >120 msec). If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility.
13. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5 × ULN,
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
14. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 3 months of Screening. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 360 mL beer, 45 mL of 40% spirit or 150 mL of wine).
15. Blood donation (excluding plasma donations) of approximately 400 mL or more within 60 days prior to dosing.
16. Participants who, in the judgment of the investigator, are not suitable for participation in the study.
17. Skin scar, rash, or ulceration at the injection site (abdomen).
18. History of vasovagal syncope or needle phobia, and inability to tolerate venous indwelling catheter blood collection.
19. Participants who plan to donate sperm or oocytes within 6 months after administration of the investigational drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events as assessed by CTCAE v5.0 | From pre-dosing to the end of follow-up at 18 weeks
  The number of AEs (e.g., abnormalities in laboratory tests, vital signs, physical examinations, and 12-lead ECGs) will be recorded and analyzed.

SECONDARY OUTCOMES:
Serum pharmacokinetics parameters (Cmax, Tmax, AUC0-inf, AUC0-t, λz, t1/2, Vz/F, and CL/F). | From pre-dosing to the end of follow-up at 18 weeks
  GB18 Serum pharmacokinetics parameters (unbound and total), including but not limited to maximum concentration (Cmax), peak time (Tmax), area under the serum concentration-time curve from time 0 to infinity (AUC0-inf), area under the serum concentration-time curve from time 0 (pre-dose) to the time t (AUC0-t), elimination rate constant (λz), elimination half-life (t1/2), apparent volume of distribution (Vz/F), apparent total serum clearance (CL/F).
Serum concentrations of total and, if feasible, unbound GDF15 specified in the schedule of activities. | From pre-dosing to the end of follow-up at 18 weeks
(if applicable) Incidence of ADA and Nab | From pre-dosing to the end of follow-up at 18 weeks

OTHER OUTCOMES:
Change from baseline of body weight at time points specified in the schedule of activities | From pre-dosing to the end of follow-up at 18 weeks
Change of QTc interval in the electrocardiogram and its correlation with the dosage of GB18 | From pre-dosing to D71 after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joo M, Kim D, Lee MW, Lee HJ, Kim JM. GDF15 Promotes Cell Growth, Migration, and Invasion in Gastric Cancer by Inducing STAT3 Activation. Int J Mol Sci. 2023 Feb 2;24(3):2925. doi: 10.3390/ijms24032925. PMID 36769245
- [Background] Tsui KH, Hsu SY, Chung LC, Lin YH, Feng TH, Lee TY, Chang PL, Juang HH. Growth differentiation factor-15: a p53- and demethylation-upregulating gene represses cell proliferation, invasion, and tumorigenesis in bladder carcinoma cells. Sci Rep. 2015 Aug 7;5:12870. doi: 10.1038/srep12870. PMID 26249737
- [Background] Lerner L, Hayes TG, Tao N, Krieger B, Feng B, Wu Z, Nicoletti R, Chiu MI, Gyuris J, Garcia JM. Plasma growth differentiation factor 15 is associated with weight loss and mortality in cancer patients. J Cachexia Sarcopenia Muscle. 2015 Dec;6(4):317-24. doi: 10.1002/jcsm.12033. Epub 2015 Apr 30. PMID 26672741
- [Background] Suzuki H, Mitsunaga S, Ikeda M, Aoyama T, Yoshizawa K, Yoshimatsu H, Kawai N, Masuda M, Miura T, Ochiai A. Clinical and Tumor Characteristics of Patients with High Serum Levels of Growth Differentiation Factor 15 in Advanced Pancreatic Cancer. Cancers (Basel). 2021 Sep 28;13(19):4842. doi: 10.3390/cancers13194842. PMID 34638326
- [Background] Niu Y, Zhang W, Shi J, Liu Y, Zhang H, Lin N, Li X, Qin L, Yang Z, Su Q. The Relationship Between Circulating Growth Differentiation Factor 15 Levels and Diabetic Retinopathy in Patients With Type 2 Diabetes. Front Endocrinol (Lausanne). 2021 Mar 15;12:627395. doi: 10.3389/fendo.2021.627395. eCollection 2021. PMID 33790859
- [Background] Siddiqui JA, Pothuraju R, Khan P, Sharma G, Muniyan S, Seshacharyulu P, Jain M, Nasser MW, Batra SK. Pathophysiological role of growth differentiation factor 15 (GDF15) in obesity, cancer, and cachexia. Cytokine Growth Factor Rev. 2022 Apr;64:71-83. doi: 10.1016/j.cytogfr.2021.11.002. Epub 2021 Nov 17. PMID 34836750
- [Background] Tsai VW, Brown DA, Breit SN. Targeting the divergent TGFbeta superfamily cytokine MIC-1/GDF15 for therapy of anorexia/cachexia syndromes. Curr Opin Support Palliat Care. 2018 Dec;12(4):404-409. doi: 10.1097/SPC.0000000000000384. PMID 30382947
- [Background] Wischhusen J, Melero I, Fridman WH. Growth/Differentiation Factor-15 (GDF-15): From Biomarker to Novel Targetable Immune Checkpoint. Front Immunol. 2020 May 19;11:951. doi: 10.3389/fimmu.2020.00951. eCollection 2020. PMID 32508832
- [Background] Grande AJ, Silva V, Sawaris Neto L, Teixeira Basmage JP, Peccin MS, Maddocks M. Exercise for cancer cachexia in adults. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD010804. doi: 10.1002/14651858.CD010804.pub3. PMID 33735441
- [Background] Balstad TR, Brunelli C, Pettersen CH, Schonberg SA, Skorpen F, Fallon M, Kaasa S, Bye A, Laird BJA, Stene GB, Solheim TS. Power Comparisons and Clinical Meaning of Outcome Measures in Assessing Treatment Effect in Cancer Cachexia: Secondary Analysis From a Randomized Pilot Multimodal Intervention Trial. Front Nutr. 2021 Jan 14;7:602775. doi: 10.3389/fnut.2020.602775. eCollection 2020. PMID 33585533
- [Background] Argiles JM, Stemmler B, Lopez-Soriano FJ, Busquets S. Inter-tissue communication in cancer cachexia. Nat Rev Endocrinol. 2018 Dec;15(1):9-20. doi: 10.1038/s41574-018-0123-0. PMID 30464312
- [Background] Ferrer M, Anthony TG, Ayres JS, Biffi G, Brown JC, Caan BJ, Cespedes Feliciano EM, Coll AP, Dunne RF, Goncalves MD, Grethlein J, Heymsfield SB, Hui S, Jamal-Hanjani M, Lam JM, Lewis DY, McCandlish D, Mustian KM, O'Rahilly S, Perrimon N, White EP, Janowitz T. Cachexia: A systemic consequence of progressive, unresolved disease. Cell. 2023 Apr 27;186(9):1824-1845. doi: 10.1016/j.cell.2023.03.028. PMID 37116469
- [Background] Yu J, Choi S, Park A, Do J, Nam D, Kim Y, Noh J, Lee KY, Maeng CH, Park KS. Bone Marrow Homeostasis Is Impaired via JAK/STAT and Glucocorticoid Signaling in Cancer Cachexia Model. Cancers (Basel). 2021 Mar 2;13(5):1059. doi: 10.3390/cancers13051059. PMID 33801569
- [Background] Naito T. Evaluation of the True Endpoint of Clinical Trials for Cancer Cachexia. Asia Pac J Oncol Nurs. 2019 Jul-Sep;6(3):227-233. doi: 10.4103/apjon.apjon_68_18. PMID 31259217
- [Background] Nishikawa H, Goto M, Fukunishi S, Asai A, Nishiguchi S, Higuchi K. Cancer Cachexia: Its Mechanism and Clinical Significance. Int J Mol Sci. 2021 Aug 6;22(16):8491. doi: 10.3390/ijms22168491. PMID 34445197
- [Background] Li Y, Jin H, Chen Y, Huang T, Mi Y, Zou Z. Cancer cachexia: molecular mechanism and pharmacological management. Biochem J. 2021 May 14;478(9):1663-1688. doi: 10.1042/BCJ20201009. PMID 33970218
- [Background] Argiles JM, Lopez-Soriano FJ, Stemmler B, Busquets S. Cancer-associated cachexia - understanding the tumour macroenvironment and microenvironment to improve management. Nat Rev Clin Oncol. 2023 Apr;20(4):250-264. doi: 10.1038/s41571-023-00734-5. Epub 2023 Feb 20. PMID 36806788
- [Background] Baazim H, Antonio-Herrera L, Bergthaler A. The interplay of immunology and cachexia in infection and cancer. Nat Rev Immunol. 2022 May;22(5):309-321. doi: 10.1038/s41577-021-00624-w. Epub 2021 Oct 4. PMID 34608281
- [Background] Evans WJ, Morley JE, Argiles J, Bales C, Baracos V, Guttridge D, Jatoi A, Kalantar-Zadeh K, Lochs H, Mantovani G, Marks D, Mitch WE, Muscaritoli M, Najand A, Ponikowski P, Rossi Fanelli F, Schambelan M, Schols A, Schuster M, Thomas D, Wolfe R, Anker SD. Cachexia: a new definition. Clin Nutr. 2008 Dec;27(6):793-9. doi: 10.1016/j.clnu.2008.06.013. Epub 2008 Aug 21. PMID 18718696